CLINICAL TRIAL: NCT04430426
Title: Heterozygous Individuals for AGXT and Kidney Stones
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kyle D. Wood, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300005327
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Kidney Stone
Keywords: kidney stone; oxalate
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled Dietary Study (Experimental): Participants will consume the controlled diet for five days and be administered an intravenous (IV) load of glycolate. Participants will provide urine and blood samples both before the glycolate load to establish baseline levels and after the glycolate load to measure oxalate levels afterwards.
  Interventions: Other: Controlled Diet; Other: Glycolate Administration

INTERVENTIONS:
Other: Controlled Diet — Participants will consume a controlled low oxalate diet for five days.
Other: Glycolate Administration — Participants will come to the UAB Clinical Research Unit (CRU) and be administered a glycolate load via intravenous (IV) catheter.

SUMMARY:
This study seeks to examine the effects of a heterozygous mutation of the AGXT gene in a stone forming population on endogenous oxalate production. Participants will consume a controlled low-oxalate diet and provide blood and urine samples to measure the amount of oxalate in their bodies. Subjects will then be administered an intravenous (IV) load of glycolate, providing additional blood and urine samples afterwards to measure any increase in oxalate levels.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* history of calcium oxalate stones
* heterozygous mutation of the AGXT gene, as evidenced by results from the Invitae Nephrolithiasis Panel
* willingness to comply with a controlled diet for five days

Exclusion Criteria:

* pregnant individuals
* individuals who are currently breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Urinary Oxalate Excretion | Baseline through Day 6
  Urinary oxalate excretion from urine samples will be measured as mg/day

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Wood, MD, Principal Investigator — University of Alabama at Birmingham